CLINICAL TRIAL: NCT02717793
Title: Comparison Between Isotonic 1 Repetition Maximum Measurement With Isometric Muscle Strength Testing In Healthy Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Manisha Parai, Lecturer, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: SERC231013
Record Dates: First submitted 2016-02-06; First posted 2016-03-24 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: No Condition, Healthy Females

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- isometric muscle strength (Experimental): isometric muscle strength was measured with a digital hand-held dynamometer. The digital hand-held dynamometer was held by the therapist against the flexor aspect of the distal forearm of the subject, on the wrist joint. Subject was asked to maintain the position and a break test was done with progressive loading of 5 seconds given by the tester. The peak isometric strength was recorded by a second tester at the end of 5 seconds. A standardised instructions and verbal encouragement was given to the subject for motivation. Subject as well as the tester was blinded to the values recorded on the digital hand-held dynamometer. An average of three measurements (with a rest period of 4 minutes in between each trial session) was recorded for the analysis. After each trial session, the rate of perceived exertion (RPE) was asked to the subject using the "1-10 Borg rating of perceived exertion scale"
  Interventions: Other: Strength testing
- 1RM measurement of muscle strength (Experimental): 1RM measurement was done using the Brzycki 1RM prediction equation. In first testing session, subject was instructed to perform a general warm up for 5 minutes. Thereafter, the subject was asked to perform 10 repetitions of the movement using the amount of resistance that the subject felt she will be able to lift for only less than 10 times. The selection of the weight is made based on a list of weights provided (1kg to 10kg). When the subject performed the movement for 10 times or more, then the resistance was increased 1kg at a time, until the subject can perform only 9 or fewer repetitions of the movement correctly throughout the range of motion. A 3 minutes rest period was given to the subject before the new attempt was done with the increased weight. A standardized verbal encouragement was provided for motivation
  Interventions: Other: Strength testing

INTERVENTIONS:
Other: Strength testing — isometric muscle strength
  1RM measurement of muscle strength

SUMMARY:
1 repetition maximum (RM) and Maximum Voluntary Contraction (MVC) with digital dynamometer are popular method of measuring muscle strength. The types of muscle contraction involved in both are different, 1RM involves isotonic muscle contraction (ITMC) and MVC with digital dynamometer involves isometric muscle contraction (IMMC). There are several risks involved in measurement of 1RM, such as delayed onset muscle soreness (DOMS) and unsafe for pathological joints etc, this can be reduced if IMMC is used in measuring strength. Though both cannot be equated as they are different type of contraction, therefore the purpose of this study was to compare between 1RM measurement and isometric MVC using a digital hand-held dynamometer in healthy females. Twenty nine young females (mean age = 20.77 ± 1.28) without any weight training experience (mean BMI = 20.43 ± 1.85) volunteered for the study. It was a crossover trial where 48 hours of rest period was given between each measurement technique. The result showed moderate correlations (r = 0.365-0.847) between 1RM and MVC. A simple linear regression analysis revealed a significant estimated regression equation for dominant and non-dominant hands. [Dominant, Y=0.391x + 1.472; Non-Dominant, Y=0.251x + 2.629; (Y: 1RM, x: Isometric)] with low standard error of estimation value of (Dominant, 0.74; Non-dominant, 0.80). The result also showed no significant difference between these derived equations and Brzycki 1RM prediction equation. Therefore, it was concluded that both prediction equations can be used interchangeably to predict the strength of a person, and thus IMMC can be used to predict 1RM in healthy females.

DETAILED DESCRIPTION:
A dynamic isotonic muscle contraction (ITMC) causes joint movement and excursion of a body segment as the muscle contracts and shortens or lengthens under tension. One repetition maximum (RM) is defined as the maximum weight a person can lift only once in a complete range of motion. It is a gold standard for measuring muscular strength therefore it is used for most of the strength training programmes. The 1RM test has been shown to be reliable in various populations. Further, setting an intensity of resistance training based on a percentage of the 1RM has been found to be effective for improving outcomes such as muscle strength, muscle power, and muscle hypertrophy. Many studies have shown increase in strength when RM testing is repeated over several days to weeks. Therefore, most testing protocols suggest that strength should be measured more than once; typically 2 or 3 testing sessions is recommended.

A familiarisation process prior to 1RM strength testing is necessary to ensure a reliable test result, this minimizes learning effect or systemic bias. It has been shown that without a familiarisation process prior to strength testing, there is a significant increase in the expression of muscle strength. In many studies, investigators have suggested that older individuals need 8-9 sessions of 1RM testing in order to increase the consistency of the 1RM measurements. Therefore, multiple familiarization sessions are beneficial for RM measurements. This draws us to a thought that such sessions may not be practical for studies examining training outcome to record the strength changes for several different resistance exercises as well as numerous other functional parameters. This unnecessarily increases the time requirement and extends the duration of the study, both of which might increase the likelihood of participant dropout in studies and loss of interest in exercise for clients. In the measure of 1RM, especially in patients, using a heavy weight and large number of repetitions imposes a greater risk of injury.

Having been said that, 1RM measurement requires a long period of testing to have a consistent value; it also requires familiarization technique which is also very intense and extensive procedure. To avoid the risk, related to the measurement of 1RM, many studies have been conducted to produce regression equations for predicting 1RM strength. There are other studies too that have been undertaken to determine the accuracy of such equations. Prediction of 1RM strength allows an exercise specialist to assess an individual's maximal lifting capacity without subjecting the novice lifter to the increased risk associated with a 1RM lift. The advantage of calculating 1RM using the formula is that, it provides the therapist with the most widely accepted measure of strength without the risks associated with the formal 1RM testing. However the 1RM load lifting also requires great concentration and considerable mental preparation for the subject which can be an extremely intense experience that leaves them unsure and scared. Although there is no real data concerning the risk of injury in this test, the potential risk may be significantly increased by using very heavy loads.

Testing 1RM uses isotonic movement which may be associated with increased risk of injury as it may include high speed of movement, inability to spread workload evenly over the entire ROM, unsafe for pathological joints, delayed onset of muscle soreness, requirement of equipment which can be expensive, and increased risk of injury, if the movement is done incorrectly. Measuring of 1 RM using the traditional way and by using prediction equation, both involve risk, therefore it brings us to an idea of the use of isometric type of movement in predicting 1RM.

Isometric contraction is a static form of exercise in which a muscle contracts and produces force without an appreciable change in the length of the muscle and without visible joint motion. It is a very popular method of testing the isometric strength of a particular muscle. It is a very easy, fast and accurate method of testing strength of a muscle. Isometric measurement by Lafayette Manual Muscle Test System (model 01163) has been proven to be highly reliable with in inter-class coefficient of 0.85. This method eliminates most of the risk factors that is observed in measuring 1 RM using the traditional way and the prediction equation. Furthermore, it is cost effective, more convenient to be done, and it does not aggravate sensitive joint surfaces. Therefore it reduces most of the risk involved in measuring 1RM using the traditional way and by using prediction equation. However, it is worth mentioning that, isometric strength measurement cannot be replaced with the 1RM measurement which is a dynamic method.

Blazevich et al in their study of reliability and validity of two isometric squat (IS) tests, reported that IS with an isometric rack showed significant and high correlation (r = 0.77) with 1RM squat. However, when Demura, S studied the relationship between 1RM and isometric measurement of squat(IS), their study showed that some component (wide stance and parallel depth) of the squat correlated well with 1 RM whereas others did not. Simple linear regression analysis in their study revealed a relationship of Y = 0.992X + 30.3 (Y: 1RM, X: IS). This suggested that the IS using a back dynamometer may become an effective index for predicting 1RM squat. However, since the standard error of an estimate provided by the regression equation was quite large, (11.19 kg) therefore, it could not estimate 1RM in non-athletes; this study concluded that estimating a 1RM by Isometric squat using a back dynamometer maybe difficult. Though some studies have been conducted to estimate 1RM from isometric strength measurement, there is a dearth in literature to prove the same. Therefore the investigators aim to find out if isometric strength can be compared with 1RM in female subjects without weight training experience. Hence the purpose of this study is to find if there can be comparisons between 1RM (Brzycki's prediction equation) measurement and isometric MVC using a digital hand-held dynamometer in healthy females.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females

Exclusion Criteria:

* musculoskeletal and neurological disorder
* history of high blood pressure
* heart disease
* rheumatologic disease that affected the mobility
* unstable cardio respiratorydisorder
* cardiovascular disorder

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1 minute after Exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Manisha, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No